CLINICAL TRIAL: NCT05925634
Title: Improving Outcomes From Cardiac Rehabilitation Among Older Adults Through Exercise Testing and Individualized Exercise Intensity Prescriptions
Brief Title: Improving Cardiac Rehabilitation Exercise Using Target Heart Rate Trial
Acronym: PACE SETTER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Collaborators: Henry Ford Hospital (Other); University of Pennsylvania (Other); Rutgers, The State University of New Jersey (Other); Springfield College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 077179
Record Dates: First submitted 2023-06-22; First posted 2023-06-29 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2024-08

CONDITIONS: Myocardial Infarction; Coronary Artery Bypass; Percutaneous Coronary Intervention; Heart Failure; Cardiac Valve Surgery
MeSH Terms: conditions — Myocardial Infarction; Heart Failure | interventions — Methods

STUDY DESIGN:
Intervention Model Description: A practical two-arm, parallel-group, open-label, efficacy randomized trial.
Who Masked: Outcomes Assessor
Masking Description: The assessment of the 6- minute walk test, handgrip strength, and Short Physical Performance Battery [SPPB]) will be performed by a blinded research team member. The blinding will occur at baseline, end of cardiac rehabilitation, and at 6 months after cardiac rehabilitation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RPE (usual care) (Active Comparator): Participants randomized to usual care (RPE) will not complete a GXT. They will instead be scheduled for an approximately 5-minute educational session (i.e., time/attention-matched control condition) where they will receive information about heart-healthy nutrition. This is standard care at both sites. Patients in the control group will follow standard exercise prescription protocols in CR. This will include a baseline exercise assessment on exercise equipment in the gym (e.g., treadmill, elliptical, rower, NuStep, and/or stationary bicycle) as appropriate. Based on exercise levels achieved on the first day, patients will be given exercise recommendations for their 2nd session of CR and so forth. Participants will be asked to exercise at a moderate intensity RPE level at both sites. As the patients progress in CR, patients will increase their time, intensity, and mode of exercise guided by RPE and clinical assessment.
  Interventions: Behavioral: RPE (usual care)
- GXT+ THHR (intervention) (Experimental): Patients assigned to the intervention group will complete a GXT approximately one week later and ideally prior to the 4th cardiac rehabilitation session. Resting and peak heart rate from the GXT will be recorded and used to calculate a target heart rate range (THRR) using the Karvonen formula (60-85% Heart rate reserve). After the test, they will receive psychoeducational feedback (PF) about their test results and exercise performance. After the PF, we will discuss the THRR and how it will be used to guide exercise intensity in CR. Patients in the intervention group will use their THHR to adjust their exercise intensity. For the first 6 cardiac rehabilitation sessions, patients will receive feedback about heart rate from the PolarHR monitor, research staff and CR staff when available. The goal is for patients to exercise in THRR for the majority of each exercise session.
  Interventions: Behavioral: GXT+THHR (intervention)

INTERVENTIONS:
Behavioral: RPE (usual care) — Patients in the active comparator group will follow standard exercise prescription protocols in cardiac rehabilitation.
  Other Names: Relative Perceived Exertion (RPE) Exercise Group
  Arms: RPE (usual care)
Behavioral: GXT+THHR (intervention) — Patients in the personalized care group will perform a graded exercise test and the peak heart rate from the test will allow the researcher to calculate a target heart rate range (THRR). Then, the patients will receive psychoeducational feedback (PF) about their test results and exercise performance. After PF, their THRR will be reviewed and how it will be used to guide exercise intensity in CR will be discussed.
  Other Names: Experimental: Graded Exercise Test (GXT) + Target Heart Rate Range (THHR)
  Arms: GXT+ THHR (intervention)

SUMMARY:
The goal of this clinical trial is to compare two types of exercise prescriptions in cardiac rehabilitation eligible older adults (60 years or older) with heart disease. The investigators found in a single site pilot trial (insert NCTxxx) that one exercise prescription was better and are now repeating this study in a larger population at two sites (Baystate Medical Center, Springfield MA and Henry Ford Health System, Detroit MI). The main questions the investigators aim to answer are:

1. Compare two different exercise prescriptions in cardiac rehabilitation on exercise outcomes

   1. Graded exercise test +Target heart rate range prescription [GXT-THRR]
   2. Rating of perceived exertion (RPE)
2. What is the role of psychological feedback on fitness outcomes during cardiac rehabilitation and physical activity outside of cardiac rehabilitation.
3. What are the long-term clinical outcomes between the two exercise prescriptions

Participants will be asked to:

* Complete surveys about physical activity, exercise anxiety, exercise efficacy, and fears about exercising
* Perform fitness measures (6-minute walk test, balance tests, stand to sit tests, a 400 meter walk, and handgrip strength)
* Attend at least 18 sessions of cardiac rehabilitation after they are randomized to their exercise prescription group
* Wear a heart rate monitor and a physical activity monitor per study protocol

Participants will be randomized (flip of a coin) to either receive a graded exercise test and psychoeducational feedback or lifestyle education (nutrition for cardiac). The graded exercise test will be used to create a personalized exercise prescription with the target heart rate range calculated from the test and the lifestyle education group will use their ratings of perceived exertion for their exercise prescription.

DETAILED DESCRIPTION:
This study aims to conduct a practical two-arm, parallel-group, open-label, efficacy randomized trial comparing Graded Exercise Testing+ Target Heart Rate Range (GXT-THRR) vs. Usual Care (UC) on changes in fitness (as measured by 6MWT, exercise training METs, handgrip strength and Short Physical Performance Battery [SPPB]) and PA behavior among 320 patients enrolled in CR. The investigators will recruit older adults (age ≥ 60 years) attending outpatient CR from two complementary but different CR centers. The investigators will compare changes in fear and self-efficacy between these two groups and measure long-term clinical outcomes. The investigators have designed the study to be as generalizable as possible, so most CR programs can immediately apply the results in clinical practice.

Eligible patients who are willing to participate will complete written informed consent. Baseline demographics, comorbidities, and prescribed medications and doses (including beta-blockers) will be collected.

Patients will then undergo a baseline assessment. This will include a 6MWT and SPPB using standard guideline procedures. During this time period, patients will also be fitted with an accelerometer to wear for 7 days (Actigraph, CenterPoint, Pensacola, FL) to assess time spent in moderate to vigorous PA (MVPA). The investigators have significant experience assessing PA, 6MWT, and SPPB, and anticipate few issues in making these measurements. Patients will also complete the following psychological assessments:

* Multidimensional Self-Efficacy for Exercise Scale. Self- efficacy is a robust predictor of exercise and PA behavior and may be influenced by exercise prescription method (GXT-THRR or UC). This validated tool will assess three dimensions of self-efficacy: task efficacy (conﬁdence in performing the elemental aspects of exercise), coping efficacy (conﬁdence in exercising under challenging circumstances), and scheduling efficacy (conﬁdence in being able to schedule regular exercise into one's lifestyle).
* Exercise Sensitivity Questionnaire (ESQ). The ESQ is an 18-item self-report measure developed by Dr. Farris that conceptualizes exercise anxiety as worry and fear about the physical sensations of exercise. The ESQ has two dimensions: (1) anxiety about cardiopulmonary sensations during exercise (i.e., blurry vision, chest pain/tightness, difficulty breathing) and (2) anxiety about pain/weakness sensations during exercise (i.e., joint/back/body pain, aches, soreness).
* Exercise Perception Questionnaire. This survey uses relevant subscales of the Intrinsic Motivation Inventory and will assess patient interest/enjoyment, as well as perceived choice, competence, pressure/tension, and effort.
* Preference for and Tolerance of Exercise Intensity Questionnaire (PRETIE-Q). This validated tool reflects a patient's general attitude towards and tolerance for higher-intensity exercise. We have included this survey as an important baseline measure, which may predict exercise gains and PA patterns.
* 36 Item Short Form Survey (SF-36). This well-validated general QOL survey has been used extensively in CR and provides a useful measure of a patient's overall physical, emotional, and social QOL.
* Fried Frailty Phenotype. This assesses physical frailty through five criteria: unintentional weight loss; weakness or poor handgrip strength; self-reported exhaustion; slow walking speed; and low physical activity.
* International Physical Activity Questionnaire-Elderly. This well-validated survey will assess levels of physical activity (moderate, moderate-vigorous, vigorous) and sedentary activity.

During the time between informed consent and randomization, patients will continue to undergo CR using UC to guide intensity. This allows for exercise-related baseline measurements to be taken, including the exercise training METs on the 3rd session of CR, as suggested by AACVPR performance measures. It also allows measurement of baseline resting HR, exercise HR, and exercise RPE.

After completing all baseline assessments (including 3 sessions of CR), patients will be randomized (1:1) to either GXT-THRR or UC. Randomization will be stratified based on age, recent cardiac surgery, and site (Baystate vs. Henry Ford.) This will be done because age may have a differential impact on exercise gains; cardiac surgery can limit the available exercise training modalities (i.e., no upper body exercises); and CR site may influence the outcome in unanticipated ways. The investigators will randomize patients through use of the Research Electronic Database Capture (REDCap) software randomization module which allows secure, sequential, and concealed group allocation, as was done in the pilot. REDCap will also be used by both sites to allow uniform data collection, capture, and entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for cardiac rehabilitation by having had a cardiac event such as a myocardial infarction (heart attack), heart failure, percutaneous coronary intervention or angioplasty with stent, coronary artery bypass graft, or heart valve surgery in the past 6 months.
* Lives in, or plans to reside in, the Springfield, MA, or greater Detroit, MI, area for the next year.
* Recruited from a Phase 2 Cardiac Rehabilitation Center at either Baystate Medical Center or Henry Ford Health System.
* Age ≥ 60 years
* Agrees to attend at least 18 sessions of cardiac rehabilitation after randomization
* Agrees to attend cardiac rehabilitation at least twice a week

Exclusion Criteria: These include conditions that alter the physiology and monitoring of resting and exercise heart rate. These also include conditions that might limit an individual's ability to exercise.

* Permanent atrial fibrillation
* Heart transplant
* Left-ventricular assist devices
* Stable angina
* High-risk un-revascularized coronary artery disease
* Symptomatic peripheral artery disease
* Aortic and/or mitral stenosis
* Any condition where exercise testing or training might be unsafe or limited

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Fitness | Baseline to final CR session
  Change in functional fitness as measured by 6 minute walk from baseline to cardiac rehabilitation (CR) completion.

SECONDARY OUTCOMES:
Training exercise workload | 3rd CR session to final CR session
  Change in metabolic equivalents of task (METs)-an objective measure of a training exercise workload as changes in scores over time and between groups.
Short Physical Performance Battery | Baseline to final CR session
  Change in Short Physical Performance Battery from baseline to final CR session
Change in functional fitness at 6 months | From end of final CR session to 6 months later.
  Change in functional fitness as measured by 6-minute walk from end of CR to 6 months later.
Change in physical performance at 6 months | From end of final CR session to 6 months later.
  Short Physical Performance Battery from end of CR to 6 months later.

OTHER OUTCOMES:
Self-efficacy (task efficacy) | Pre-Post GXT
  Acute change in self-efficacy (task efficacy) measured before and after the intervention (graded exercise test (GXT) vs. time matched control) will be assessed via the Multidimensional Self-Efficacy for Exercise Scale as changes in scores over time and between groups.
Fear of Exercise | Pre-Post GXT
  Acute effects of GXT vs. time matched control on fear will be measured via the Exercise Sensitivity Questionnaire as changes in scores over time and between groups.
Reassurance | Pre-Post GXT
  Acute effects of GXT on reassurance will be measured via the Reassurance Scale as change scores over time and between groups.
Exercise Anxiety | Baseline to final CR session
  Change in exercise anxiety from baseline to final CR session over time and between groups will be measured via the Exercise Sensitivity Questionnaire.
Exercise Self-Efficacy | Baseline to final CR session
  Change in exercise self-efficacy from baseline to final CR session over time and between groups will be measured via the Preference for and Tolerance of Exercise Intensity Questionnaire.
Task Efficacy | Baseline to final CR session
  Change in task self-efficacy from baseline to final CR session over time and between groups will be measured via the Multidimensional Self-Efficacy for Exercise Scale.
Change in Quality of Life | Baseline to final CR session
  Change in Quality of Life measured by the SF-36 from baseline to the end of CR
Change in 7-day % time in Moderate to Vigorous Physical Activity | Baseline to final CR session
  Total minutes/day in moderate to vigorous physical activity that is structured exercise behavior measured with an accelerometer.
Self-reported moderate to vigorous physical activity (MVPA) over the past 7 days | Baseline to CR end, and at 3 and 6 months post CR
  Using the International physical activity questionnaire (IPAQ) to measure self-reported moderate to vigorous physical activity (MVPA) over the past 7 days
Major adverse cardiac event (death, myocardial infarction, stroke) | At end of CR up to 2 years follow-up
  A cardiovascular event including myocardial infarction or stroke, or death via reporting of events in the follow-up surveys via REDCap links or phone calls.
Admission to the hospital (full admission or observation status) with apparent life-threatening illness | At end of CR up to 2 years follow-up
  Any full admission or observation status admission to a hospital with apparent life-threatening illness via reporting of events in the follow-up surveys via REDCap links or phone calls.
Clinically indicated ischemic evaluation (exercise stress test, nuclear stress test, exercise echo, cardiac catheterization) | At end of CR up to 2 years follow-up
  A clinically indicated ischemic event during exercise stress test, nuclear stress test, exercise echo or cardiac catheterization via reporting of events in the follow-up surveys via REDCap links or phone calls.
Number of sessions of CR completed (maximum of 36) within 6 months of enrollment. | Start to end of CR
  After enrollment to cardiac rehabilitation (CR) the number of sessions completed within 6 months, with a maximum of 36 possible via the case report forms completed per participant.

CONTACTS AND LOCATIONS:
Overall Officials: Quinn R Pack, MD, Principal Investigator — Baystate Medical Center
Locations (2):
- United States (2):
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Health System, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No